CLINICAL TRIAL: NCT02849639
Title: INtervention for Cognitive Reserve Enhancement in Delaying the Onset of Alzheimer's Symptomatic Expression: The INCREASE Study
Brief Title: The INCREASE Study - Delaying the Onset of Alzheimer's Symptomatic Expression
Acronym: INCREASE
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Daniela Moga (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor-Investigator, Daniela Moga, Sponsor/PI, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 16-0375-F2L INCREASE; 1R01AG054130-01 (NIH)
Record Dates: First submitted 2016-07-15; First posted 2016-07-29 (Estimated); Results first posted 2022-08-22 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2023-06

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: deprescribing; medication therapy management
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — Medication Therapy Management; Methods

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Participants enrolled into this arm will only receive educational materials, but will not receive specific recommendations to make changes to the medications they are taking.
  Cognitive testing at the beginning and the end of the study will be done with and without a scopolamine patch to reveal cognitive reserve.
  Interventions: Other: Placebo; Drug: Scopolamine patch
- Medication Therapy Management (MTM) (Active Comparator): Participants enrolled into this arm will receive educational materials and will have their medications assessed; recommendations for changes in the medications taken will be made when appropriate.
  Cognitive testing at the beginning and the end of the study will be done with and without a scopolamine patch to reveal cognitive reserve.
  Interventions: Other: Medication Therapy Management (MTM); Drug: Scopolamine patch

INTERVENTIONS:
Other: Placebo — Participants will receive educational materials, but will not receive MTM.
  Other Names: Control
  Arms: Placebo
Other: Medication Therapy Management (MTM) — Participants will receive MTM in addition to the educational materials.
  Other Names: Intervention
  Arms: Medication Therapy Management (MTM)
Drug: Scopolamine patch — At the beginning and end of the study, participants will be asked to use a scopolamine patch. This patch is not being used to prevent motion sickness (as approved by the FDA), but instead is being used to challenge the participant's memory and thinking abilities and determine cognitive reserve.
  Other Names: Scopolamine Challenge

SUMMARY:
The study will examine the impact on cognitive reserve of a pharmacist-physician patient-centered medication therapy management intervention to address inappropriate medication use as identified by the Beers 2015 list. By bolstering cognitive reserve, this project will directly address the National Alzheimer's Project Act 2015 priorities serving to delay onset of symptoms in preclinical dementia. The results of this study will provide valuable insights on how to expand this intervention to reduce the prevalence and associated healthcare costs of symptomatic Alzheimer's disease.

DETAILED DESCRIPTION:
This is a 12-month, parallel arm, study to be conducted at the University of Kentucky. The study will involve assessing medication use and identifying any medicines that may be inappropriate for elderly adults.

At the beginning of the study, participants will be asked to undergo one amyloid-PET scan to detect early amyloid plaques in their brain which could increase the risk of Alzheimer's disease in the near future. In addition, at the beginning and end of the study, participants will be asked to use a scopolamine patch. This patch is not being used to prevent motion sickness (as approved by the FDA), but instead is being used to challenge the participant's memory and thinking abilities.

Part of the study includes collecting information regarding participants memory and thinking abilities. Participants will be asked to complete questionnaires as well as memory and thinking tests.

A study doctor will review participants medical history and then perform routine medical (physical and neurological) examinations.

Two of the study visits will be conducted by phone to check up on the participants.

At the beginning, middle, and end of the study, participants will meet with a doctor and pharmacist to review and make any changes deemed appropriate to their current medicines. This will be done in order to try and eliminate medicines that are not recommended for the elderly. These visits are referred to as the Medication Therapy Management (MTM).

ELIGIBILITY:
Inclusion Criteria:

* Non-demented
* No previous reaction or contraindication to scopolamine patch, or medical condition warranting dose adjustment in scopolamine including but not limited to: open angle glaucoma, gastrointestinal or urinary outlet obstructions, seizures, or psychosis.
* No contraindications to Aβ-PET scan including hypersensitivity to PET ligand or radiation exposures in the past year that would exceed the acceptable safe annual exposure in combination with the Aβ PET
* Medically stable and able to complete all study activities, as determined by the investigator
* Reporting at least one potentially inappropriate medication as listed in the Beers 2015 criteria
* Living in the community
* Willing to participate in this intervention study

Exclusion Criteria:

* Allergy or other know intolerance to scopolamine patches
* Narrow-angle glaucoma
* Difficulty swallowing
* Stomach or bowel problems (e.g., blockage, muscle weakness, ulcerative colitis)
* Bleeding
* Acid reflux disease
* Myasthenia gravis
* Blockage of the urinary tract.
* Seizures
* Psychosis

Ages: 65 Years to 101 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 90 (Actual)
Dates: Start 2017-04-04 (Actual); Primary Completion 2021-04-21 (Actual); Study Completion 2021-04-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Daniela Moga, MD, PhD, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Moga DC, Beech BF, Abner EL, Schmitt FA, El Khouli RH, Martinez AI, Eckmann L, Huffmyer M, George R, Jicha GA. INtervention for Cognitive Reserve Enhancement in delaying the onset of Alzheimer's Symptomatic Expression (INCREASE), a randomized controlled trial: rationale, study design, and protocol. Trials. 2019 Dec 30;20(1):806. doi: 10.1186/s13063-019-3993-0. PMID 31888732
- [Result] Moga DC, Abner EL, Schmitt FA, Eckmann L, Huffmyer M, Martinez AI, Beech BF, George R, El Khouli RH, Ali D, Jicha GA. Intervention for Cognitive Reserve Enhancement in Delaying the Onset of Alzheimer's Symptomatic Expression (INCREASE) Study: Results from a Randomized Controlled Study of Medication Therapy Management Targeting a Delay in Prodromal Dementia Symptom Progression. J Prev Alzheimers Dis. 2022;9(4):646-654. doi: 10.14283/jpad.2022.55. PMID 36281668
- [Derived] Smith NI, Martinez AI, Huffmyer M, Eckmann L, George R, Abner EL, Jicha GA, Moga DC. Acceptability of patient-centered, multi-disciplinary medication therapy management recommendations: results from the INCREASE randomized study. BMC Geriatr. 2023 Mar 10;23(1):137. doi: 10.1186/s12877-023-03876-4. PMID 36894900

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Participants enrolled into this arm will only receive educational materials, but will not receive specific recommendations to make changes to the medications they are taking.
  Cognitive testing at the beginning and the end of the study will be done with and without a scopolamine patch to reveal cognitive reserve.
  Placebo: Participants will receive educational materials, but will not receive MTM.
  Scopolamine patch: At the beginning and end of the study, participants will be asked to use a scopolamine patch. This patch is not being used to prevent motion sickness (as approved by the FDA), but instead is being used to challenge the participant's memory and thinking abilities and determine cognitive reserve.
- Medication Therapy Management (MTM): Participants enrolled into this arm will receive educational materials and will have their medications assessed; recommendations for changes in the medications taken will be made when appropriate.
  Cognitive testing at the beginning and the end of the study will be done with and without a scopolamine patch to reveal cognitive reserve.
  Medication Therapy Management (MTM): Participants will receive MTM in addition to the educational materials.
  Scopolamine patch: At the beginning and end of the study, participants will be asked to use a scopolamine patch. This patch is not being used to prevent motion sickness (as approved by the FDA), but instead is being used to challenge the participant's memory and thinking abilities and determine cognitive reserve.
Period: Overall Study
Arm/Group | Placebo | Medication Therapy Management (MTM)
Started | 44 | 46
Completed | 41 | 44
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Medication Therapy Management (MTM) | Total
Number analyzed (Participants) | 44 | 46 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 74.1 (6.6) | 73.4 (5.6) | 73.9 (6.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 34 | 57
  Male | 21 | 12 | 33
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 44 | 46 | 90
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 2 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 6 | 8
  White | 40 | 40 | 80
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Standardized Uptake Value ratio [Count of Participants; unit: Participants] — Quantitative SUVR determinations based on Aβ-PET imaging allow for the specification of amyloid burden as a continuous variable. We used predefined cut-off points at 1.2 and 1.4 to categorize amyloid burden. Values grater than 1.4 in the absence of cognitive impairment indicate a preclinical Alzheimer's Disease state.
  Participants
    SUVr<1.2 | 13 | 14 | 27
    1.2<=SUVr<1.4 | 17 | 17 | 34
    SUVr>=1.4 | 14 | 15 | 29
Years of education [Mean (Standard Deviation); unit: years] | 16.4 (2.6) | 16.5 (3.0) | 16.5 (2.8)
Total number of medications [Mean (Standard Deviation); unit: medications] | 12.9 (4.8) | 12.7 (5.0) | 12.8 (4.8)
Number of medications on 2015 Beers list [Mean (Standard Deviation); unit: medications] — Beers criteria list medications that are considered potentially inappropriate for adults 65 years and older. The list is updated on a regular basis through expert panel review under the American Geriatrics Society.
  medications | 2.2 (1.2) | 2.5 (1.2) | 2.4 (1.2)
Medication appropriateness index [Mean (Standard Deviation); unit: units on a scale] — The MAI rates medications as "appropriate", "marginally appropriate", or "inappropriate" based on ten criteria. All medications reported by study participants were evaluated by the study team and assigned a medication-specific MAI. As an outcome measure, the total MAI was obtained by adding the medication specific MAIs for all medications reported by the participant. Minimum score for one medication is 0 (appropriate) and the maximum is 18 (inappropriate for all criteria). Total MAI depends on the number of medications taken by participant.
  units on a scale | 10.6 (7.4) | 13.5 (9.4) | 12.1 (8.5)

OUTCOME MEASURES:

1. Primary Outcome: Medication Appropriateness Index
Description: Change from baseline to end of study. The Medication Appropriateness Index (MAI) rates medications as "appropriate", "marginally appropriate", or "inappropriate" based on ten criteria. All medications reported by study participants were evaluated by the study team and assigned a medication-specific MAI. As an outcome measure, the total MAI was obtained by adding the medication specific MAIs for all medications reported by the participant. Minimum score for one medication is 0 (appropriate) and the maximum is 18 (inappropriate for all criteria). Total MAI depends on the number of medications taken by participant. A decrease in MAI from baseline to end of study indicates improvement in medication appropriateness.
Time Frame: change from baseline to end of study, an average of 1 year
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Placebo | Medication Therapy Management (MTM)
Number analyzed (Participants) | 41 | 44
units on a scale | 11.2 (0.6) | 9.4 (0.6)

2. Primary Outcome: Trail Making Test B With the Scopolamine Patch
Description: End of study for Trail Making Test B with the scopolamine patch. The mean and standard used to compute the TMTB z-scores were taken from a sample of cognitively intact older adult research volunteers (Weintraub et al. 2009; mean = 90.3, SD = 50) (22). Z-scores were then multiplied by -1 to facilitate interpretation, since higher TMTB scores are worse. For the z-score, we converted time in seconds to units of standard deviations from a mean of 0, where 0 represents the mean performance of cognitively intact (normal) older adult research volunteers enrolled in longitudinal studies at Alzheimer's Disease Research Centers in the United States. Scores that are at least 1.5 standard deviations below the mean are indicative of potential cognitive impairment.
Time Frame: baseline to end of study, an average of 1 year
Measure: Least Squares Mean (Standard Error); unit: z-scores
Arm/Group | Placebo | Medication Therapy Management (MTM)
Number analyzed (Participants) | 40 | 42
z-scores | -0.1 (0.14) | 0.03 (0.14)

3. Secondary Outcome: Cognitive Reserve: Montreal Cognitive Assessment
Description: Change from baseline to end of study for Montreal Cognitive Assessment. Z score is based on the NACC cognitively normal population (https://files.alz.washington.edu/documentation/weintraub-2018-v3.pdf), Z score = 0 corresponds mean MoCA score for cognitively normal older adults; higher Z scores are better; typical neuropsych interpretation of z scores is that -1.5 indicates impaired performance on that test.
Time Frame: change from baseline to end of study, an average of 1 year
Population: MoCA (Z score, NACC UDS norms), challenged condition
Measure: Least Squares Mean (Standard Error); unit: z-score
Groups:
- Placebo: Participants enrolled into this arm will only receive educational materials
- Medication Therapy Management (MTM): Participants enrolled into this arm will receive educational materials and will have their medications assessed; recommendations for changes in the medications taken will be made when appropriate
Arm/Group | Placebo | Medication Therapy Management (MTM)
Number analyzed (Participants) | 41 | 44
z-score | -0.15 (0.12) | -0.31 (0.13)

4. Secondary Outcome: Cognitive Reserve: California Verbal Learning Test
Description: Change from baseline to end of study for California Verbal Learning test. Z scores (higher scores are better; Z score = 0 corresponds mean CVLT score for cognitively normal older adults; typical neuropsych interpretation of z scores is that -1.5 indicates impaired performance on that test) are adjusted for age and sex and are based on the normative population used to develop norms for CVLT-II; "individuals sampled to create the normative data were tested cross-sectionally, demographically matched to the most recent U.S. Censuses, and screened for self-reported neurological, psychiatric, or debilitating medical illnesses." Delis, D. C., Kramer, J. H., Kaplan, E., & Ober, B. A. (1987-2000). California Verbal Learning Test--Second Edition (CVLT -II) [Database record]. APA PsycTests.
  https://doi.org/10.1037/t15072-000
Time Frame: change from baseline to end of study, an average of 1 year
Population: CVLT Long Delay (Z score), challenged condition
Measure: Least Squares Mean (Standard Error); unit: z-score
Arm/Group | Placebo | Medication Therapy Management (MTM)
Number analyzed (Participants) | 41 | 44
z-score | -0.10 (0.15) | -0.083 (0.14)

5. Secondary Outcome: Perceived Health Status
Description: Change from baseline to end of study for Short Form Health Survey (SF-36). T scores have a mean of 50 and SD of 10; higher scores are better; mean = 50 represents expected mean in general US adult population, with no available clinically relevant thresholds .
Time Frame: change from baseline to end of study, an average of 1 year
Population: SF-36 Mental Component Score (T score), challenged condition
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Placebo | Medication Therapy Management (MTM)
Number analyzed (Participants) | 41 | 44
t-score | 41.4 (1.2) | 41.2 (1.3)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Placebo | Medication Therapy Management (MTM)
All-Cause Mortality (participants affected / at risk) | 2/44 | 0/46
Serious Adverse Events (participants affected / at risk) | 9/44 | 7/46
Other Adverse Events (participants affected / at risk) | 42/44 | 41/46
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Medication Therapy Management (MTM) (N=46)
Injurious fall (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Infections (Infections and infestations) | 1 (1) | 4 (4)
Major cardiac event (Cardiac disorders) | 2 (2) | 1 (1)
Stroke (Vascular disorders) | 1 (1) | 1 (1)
GI emergencies (Gastrointestinal disorders) | 2 (2) | 1 (1)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Surgical complications (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Car accident (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=44) | Medication Therapy Management (MTM) (N=46)
Neurological (Nervous system disorders) | 28 (32) | 29 (34)
GI (Gastrointestinal disorders) | 24 (26) | 27 (27)
Infections (Infections and infestations) | 9 (9) | 7 (8)
Allergies (Immune system disorders) | 1 (1) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 16 (16) | 21 (22)
Cardiovascular (Cardiac disorders) | 6 (6) | 5 (5)
Renal and GU (Renal and urinary disorders) | 3 (4) | 3 (3)
Skin (Skin and subcutaneous tissue disorders) | 3 (3) | 5 (5)
Other (General disorders) | 3 (3) | 3 (3)
Metabolic (Metabolism and nutrition disorders) | 5 (5) | 5 (6)
Visual (Eye disorders) | 3 (3) | 5 (5)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Auditory (Ear and labyrinth disorders) | 2 (2) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-02-27): https://cdn.clinicaltrials.gov/large-docs/39/NCT02849639/Prot_001.pdf
  • Statistical Analysis Plan (2015-12-14): https://cdn.clinicaltrials.gov/large-docs/39/NCT02849639/SAP_002.pdf
  • Informed Consent Form (2019-11-20): https://cdn.clinicaltrials.gov/large-docs/39/NCT02849639/ICF_000.pdf